CLINICAL TRIAL: NCT03862482
Title: Prospective Randomised Clinical Trial Evaluating the Effects of Two Different Implant Collar Designs on Peri-Implant Healing and Functional Osseointegration After 25 Years of Function With Full Arch Mandibular Prostheses
Brief Title: Peri-Implant Healing Around Two Different Machined-Collar Designs After 25 Years of Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Aldo Joseph Camarda, Principal Investigator, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CERC-19-015-P
Record Dates: First submitted 2019-02-20; First posted 2019-03-05 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Jaw, Edentulous
Keywords: Dental Implants, Microtextured Fixture, Machined Collar
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: For the initial study, a statistician had prepared a sampling design that included three configuration diagrams. Each diagram identified five implants of the three types, and showed how one of each type was to be placed in a cyclical, side-by-side, rotating fashion at five sites between mental foramena. Allocation concealment by the project coordinator then allowed 20 participants to receive Configuration 1, 19 had Configuration 2, and 19 had Configuration 3. Configuration diagram (but not number) was stored inside each chart, and only shown to the operating team at the time of surgery.
  The present study is a continuation of this clinical trial, including data collected at the 25-year (24.6 ± 0.19 years, mean ± SE) follow-up. Twenty-two of the original participants (41.5%, age 71.1 ± 1.2 years, 11 women, 110 implants) were enrolled in this study. Eight participants (40 implants) received Configuration 1, 8 (40 implants) had Configuration 2, and 6 (30 implants) had Configuration 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1 (Configuration 1) (Active Comparator): Device placement: B (Brånemark® dental implant) placed at two sites, SW (Swede-Vent® dental implant) placed at two sites, SC (Screw-Vent® dental implant) placed at one site
  Interventions: Device: Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1 (Configuration 1)
- Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2 (Configuration 2) (Experimental): Device placement: B (Brånemark® dental implant) placed at one site, SW (Swede-Vent® dental implant) placed at two sites, SC (Screw-Vent® dental implant) placed at two sites
  Interventions: Device: Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2 (Configuration 2)
- Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3) (Experimental): Device placement: B (Brånemark® dental implant) placed at two sites, SW (Swede-Vent® dental implant) placed at one site, SC (Screw-Vent® dental implant) placed at two sites
  Interventions: Device: Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3)

INTERVENTIONS:
Device: Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1 (Configuration 1) — Brånemark® implant placed at sites 2 (left medial) and 5 (right distal), Swede-Vent® implant placed at sites 1 (left distal) and 4 (right medial), Screw-Vent® implant placed at site 3 (para symphysis)
  Arms: Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1 (Configuration 1)
Device: Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2 (Configuration 2) — Brånemark® implant placed at site 3 (para symphysis), Swede-Vent® implant placed at sites 2 (left medial) and 5 (right distal), Screw-Vent® implant placed at sites 1 (left distal) and 4 (right medial)
  Arms: Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2 (Configuration 2)
Device: Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3) — Brånemark® implant placed at sites 1 (left distal) and 4 (right medial), Swede-Vent® implant placed at site 3 (para symphysis), Screw-Vent® implant placed at sites 2 (left medial) and 5 (right distal)
  Arms: Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3)

SUMMARY:
Brånemark System® dental implant osseointegration was introduced in 1965 as a novel approach to the replacement of missing teeth. Although this implant's machined, screw-shaped surface had excellent, well-documented, short- and long-term clinical success (Adell, R. 1987; Albrektsson, T., et al., 1981; Albrektsson, T., et al., 1986; Brånemark, P-I. , 1983; Brånemark P-I. 1987), newer implant designs were introduced that could enhance fusion of the implant to jaw bones, and better resist functional forces. One such implant, Screw-Vent®, has a fixture macro structure very similar to that of the Brånemark® implant. However, its fixture surface was acid etched (1-3µm) which could enhance osseointegration, and it has a longer, narrower machined internal-hex, friction-fit collar that could better resist functional forces.These characteristics should lead to less bone loss (Niznick, G. A., 1989). However, one clinical study (De Bruyen, et al., 1992) reported greater short-term bone loss with this implant compared to the Brånemark® implant, possibly due to its longer machined collar, and advocated long-term clinical studies. Therefore, this prospective within-subject clinical trial was undertaken in 1993 to first compare the Brånemark® implant with another implant, Swede-Vent®, a copy of the Brånemark® macro structure except for its fixture surface that was identically micro textured as that of Screw-Vent® by the same manufacturer. The effect on bone healing could then be compared between Brånemark®'s machined and Swede-Vent®'s micro textured fixture surfaces in the short- and long-terms. Since Screw-Vent®'s fixture surface was identically micro textured as that of Swede-Vent®, the investigators could then evaluate and compare the effects on bone healing of Screw-Vent®'s longer, narrower, internal-connection machined collar to the identical shorter, wider, external-connection machined collars of the Swede-Vent® and Brånemark® implants. All three two-part, platform-matched, parallel-wall implants were made of commercially pure titanium, had a very similar fixture macro design, were approved by the Food and Drug Administration (USA) and Health and Welfare Canada, and were commercially available in North America. Brånemark® and Screw-Vent® implants are still available, but the Swede-Vent® implant is not.

DETAILED DESCRIPTION:
Therefore, between 1993 and 1996, 58 of 60 eligible participants had been recruited into a prospective, randomized clinical trial. This trial had been peer reviewed, had received ethical approval, and had taken place at the Université de Montréal's Faculty of Dental Medicine and its affiliated hospital dental department. Follow-up documentation occurred at one year, two years, and 15 to 20 years following prostheses attachment (ClinicalTrials Identification Number NCT01641198), and the results were published (Camarda, et al., 2018). The present study reports on data collected at the 25-year (24.6 ± 0.19 years, mean ± SE) follow-up (ClinicalTrials Identification Number NCT03862482), focusing specifically on the evaluation and comparison of the effects on peri-implant healing and functional osseointegration of the two different machined collar designs. That is to say, the identical shorter, wider, external-connection Brånemark® and Swede-Vent® collars versus the longer, narrower, internal-connection Screw-Vent® collar. Twenty-two of the original participants (41.5%, age 71.1 ± 1.2 years, 11 women, 110 implants) were enrolled into this study. All study procedures were performed in accordance with the Helsinki Declaration and its later amendments, and all participants signed informed consent documents prior to inclusion into this study.

ELIGIBILITY:
Inclusion Criteria:

* non-smoker
* no temporomandibular joint (TMJ) disorder or facial pain
* having participated in the original study (1993 - 1996) at which time the minimum participants' age was 25 years and the maximum 56 years

Exclusion Criteria:

* refusal to sign informed consent documents

Ages: 48 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aldo J Camarda, DDS, MSc, Principal Investigator — Université de Montréal; Robert Durand, DMD, MSc, Principal Investigator — Université de Montréal; Marwa Benkarim, Principal Investigator — Université de Montréal; Pierre Rompré, MSc, Principal Investigator — Université de Montréal; Geneviève Guertin, DMD, MSc, Principal Investigator — Université de Montréal; Hugo Ciaburro, DMD, MSc, Study Director — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adell, R. (1987). Long-term treatment results. In: Brånemark, P-I., Zarb, G.A., Albrektsson, T. (Eds.). Tissue-integrated prostheses: osseointegration in clinical dentistry (pp. 175-285). Quintessence Publishing Co. Inc.
- [Background] Albrektsson T, Branemark PI, Hansson HA, Lindstrom J. Osseointegrated titanium implants. Requirements for ensuring a long-lasting, direct bone-to-implant anchorage in man. Acta Orthop Scand. 1981;52(2):155-70. doi: 10.3109/17453678108991776. PMID 7246093
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Bhaskaran V, Qualtrough AJ, Rushton VE, Worthington HV, Horner K. A laboratory comparison of three imaging systems for image quality and radiation exposure characteristics. Int Endod J. 2005 Sep;38(9):645-52. doi: 10.1111/j.1365-2591.2005.00998.x. PMID 16104978
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Branemark PI. Osseointegration and its experimental background. J Prosthet Dent. 1983 Sep;50(3):399-410. doi: 10.1016/s0022-3913(83)80101-2. No abstract available. PMID 6352924
- [Background] Brånemark P-I. (1987). Introduction to osseointegration. In Brånemark, P-I., Zarb, G.A., Albrektsson, T. (Eds.). Tissue-integrated prostheses: osseointegration in clinical dentistry (pp. 11-76). Quintessence Publishing Co. Inc.
- [Background] De Bruyn H, Collaert B, Linden U, Flygare L. A comparative study of the clinical efficacy of Screw Vent implants versus Branemark fixtures, installed in a periodontal clinic. Clin Oral Implants Res. 1992 Mar;3(1):32-41. doi: 10.1034/j.1600-0501.1992.030106.x. PMID 1420725
- [Background] Galgut P. A comparison of different indices used in the clinical assessment of plaque and gingival bleeding. Clin Oral Investig. 1999 Jun;3(2):96-9. doi: 10.1007/s007840050085. PMID 10803118
- [Background] Niznick, G. A. (1989). Open letters no. 1 and no. 2 to the dental profession, Core-Vent Corporation Newsletter and manufacturer's product description. Encino, California USA.
- [Result] Camarda AJ, Durand R, Benkarim M, Rompre PH, Guertin G, Ciaburro H. Prospective randomized clinical trial evaluating the effects of two different implant collar designs on peri-implant healing and functional osseointegration after 25 years. Clin Oral Implants Res. 2021 Mar;32(3):285-296. doi: 10.1111/clr.13699. Epub 2021 Jan 25. PMID 33314332
- [Result] Camarda AJ, Milot P, Ciaburro H, Rompre PH, Sallaleh I, Do CMA. Long-term randomized clinical trial evaluating the effects of fixture surface acid-etching and machined collar design on bone healing. Quintessence Int. 2018;49(9):733-743. doi: 10.3290/j.qi.a41013. PMID 30202836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment date: May 1st - May 30th, 2019. Recruitment location: Faculty of Dental Medicine
Units Other Than Participants: Implants
Groups:
- Active Comparator: Brånemark® (B) 2, Swede-Vent® (SW) 2, Screw-Vent® (SC) 1 (Configuration 1): Device: Brånemark® implant placed at sites 2 (left medial) and 5 (right distal), Swede-Vent® implant placed at sites 1 (left distal) and 4 (right medial), Screw-Vent® implant placed at site 3 (para symphysis) between mandibular foramen
- Experimental: Brånemark® (B) 1, Swede-Vent® (SW) 2, Screw-Vent® (SC) 2 (Configuration 2): Device: Brånemark® implant placed at site 3 (para symphysis), Swede-Vent® implant placed at sites 2 (left medial) and 5 (right distal), Screw-Vent® implant placed at sites 1 (left distal) and 4 (right medial) between mandibular foramen
- Experimental: Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3): Device: Brånemark® implant placed at sites 1 (left distal) and 4 (right medial), Swede-Vent® implant placed at site 3 (para symphysis), Screw-Vent® implant placed at sites 2 (left medial) and 5 (right distal) between mandibular foramen
Period: Overall Study
Arm/Group | Active Comparator: Brånemark® (B) 2, Swede-Vent® (SW) 2, Screw-Vent® (SC) 1 (Configuration 1) | Experimental: Brånemark® (B) 1, Swede-Vent® (SW) 2, Screw-Vent® (SC) 2 (Configuration 2) | Experimental: Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3)
Started | 8; 40 Implants (Eight participants (forty implant units) were randomly allocated to Configuration 1 by study coordinator. Each participant was also randomly assigned one of the three implant units (B or SW or SC) on a rotating basis to one of five sites between mental foramen. As a result, an equal number of each implant unit type was placed at each the five sites) | 8; 40 Implants (Eight participants (forty implant units) were randomly allocated to Configuration 2 by study coordinator. Each participant was also randomly assigned one of the three implant units (B or SW or SC) on a rotating basis to one of five sites between mental foramen. As a result, an equal number of each implant unit type was placed at each the five sites) | 6; 30 Implants (Six participants (thirty implant units) were randomly allocated to Configuration 3 by study coordinator. Each participant was also randomly assigned one of the three implant units (B or SW or SC) on a rotating basis to one of five sites between mental foramen. As a result, an equal number of each implant unit type was placed at each the five sites)
Completed | 8; 39 Implants (Sixteen B, 16 SW, and eight SC implant units were placed on a rotating basis at the five sites for a total of 40 implant units. Of these, one implant unit (SW) had fractured and was subsequently excluded from all future analyses) | 8; 38 Implants (Eight B, 16 SW, and 16 SC implant units were placed on a rotating basis at the five sites for a total of 40 implant units. Of these, two implant units (one B, one SW) were removed from all future analyses due to technical issues with radiographs) | 6; 30 Implants (Twelve B, six SW, and 12 SC implant units were placed on a rotating basis at the five sites for a total of 30 implant units)
Not Completed | 0; 1 Implants | 0; 2 Implants | 0; 0 Implants

BASELINE CHARACTERISTICS:
Population: Each of the total 22 participants contributed five units (implants) for a total of 110 implants (B=36, SW=38, SC=36).
Units Other Than Participants: Implants
Groups:
- Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1 (Configuration 1): Device placement: B (Brånemark® dental implant unit) placed at sites 2 (left medial) and 5 (right distal), SW (Swede-Vent® dental implant unit) placed at sites 1 (left distal) and 4 (right medial), SC (Screw-Vent® dental implant unit) placed at site 3 (para symphysis) for a total of 40 dental implant units (16 B, 16 SW, 8 SC), all between mandibular foramen
- Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2 (Configuration 2): Device placement: B (Brånemark® dental implant unit) placed at site 3 (para symphysis), SW (Swede-Vent® dental implant unit) placed at sites 2 (left medial) and 5 (right distal), SC (Screw-Vent® dental implant unit) placed at sites 1 (left distal) and 4 (right medial) for a total of 40 dental implant units (eight B, 16 SW, 16 SC), all between mandibular foramen
- Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3): Device placement: B (Brånemark® dental implant unit) placed at sites 1 (left distal) and 4 (right medial), SW (Swede-Vent® dental implant unit) placed at site 3 (para symphysis), SC (Screw-Vent® dental implant unit) placed at sites 2 (left medial) and 5 (right distal) for a total of 30 dental implant units (12 B, six SW, 12 SC), all between mandibular foramen
- Total: Total of all reporting groups
Arm/Group | Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1 (Configuration 1) | Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2 (Configuration 2) | Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3) | Total
Number analyzed (Participants) | 8 | 8 | 6 | 22
Number analyzed (Implants) | 40 | 40 | 30 | 110
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (Years): Mean ± Standard Deviation | 69.4 (6.12) | 71.5 (5.09) | 70.5 (4.11) | 70.45 (5.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of Men and Women for each Configuration.
  Participants
    Female | 4 | 5 | 2 | 11
    Male | 4 | 3 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 6 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Total number of implant units per study arm [Number; unit: Number count] — Count of total number of implant units per study arm entered into study at baseline
  Number count | 40 | 40 | 30 | 110

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Distance Between First Bone to Implant Contact Point (fBIC) and Microgap (MG), After 25 Years of Function, Between All B, All SW, and All SC Dental Implant Units in All Three Configurations
Description: Distance between first bone-to-implant contact point (fBIC) and microgap (MG) at the crest was measured (mm) at mesial and distal sides of each implant/abutment complex on conventional peri-apical radiographs using a standardized equipment and measurement protocol (Camarda, et al., 2018) after 25 years of function. Values fBIC-MG (Mean ± SE) ("-" for bone loss) were calculated, recorded and compared between all B and all SW, between all B and all SC and between all SW and all SC dental implant units in all three Configurations
Time Frame: After 25 years (24.6 ± 0.19 years, mean ± SE) of function
Population: 22 participants in all Configurations contributed 110 implant units (40 Configuration 1, 40 Configuration 2, and 30 Configuration 3). One implant unit (SW, Configuration 1) had fractured, and two implant units (B and SW, Configuration 2) were excluded due to technical difficulties with radiographic technique. Consequently, 107 implant units were were analyzed.
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: Implants
Groups:
- All Participants (Configurations 1, 2, and 3): Configuration 1: Device placement: B (Brånemark® dental implant unit) placed at sites 2 (left medial) and 5 (right distal)
  Configuration 2: Device placement SW (Swede-Vent® dental implant unit) placed at sites 2 (left medial) and 5 (right distal)
  Configuration 3: Device placement SC (Screw-Vent® dental implant unit) placed at sites 2 (left medial) and 5 (right distal)
Arm/Group | All Participants (Configurations 1, 2, and 3)
Number analyzed (Participants) | 22
Number analyzed (Implants) | 107
mm
  Total 35 Brånemark® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 35
  Total 35 Brånemark® dental implant units analyzed for all three Configurations | -0.85 (0.18)
  Total 36 Swede-Vent® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 36
  Total 36 Swede-Vent® dental implant units analyzed for all three Configurations | -1.00 (0.18)
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 36
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations | -1.77 (0.18)
Statistical Analysis 1: Comparison: All Participants (Configurations 1, 2, and 3); Total 35 Brånemark® implants analyzed for all Configurations. Size difference expected 0.95 bone level change between B/SW/SC. Sample size 16 participants ensured 80% power to reject null hypothesis (two-sided Bonferroni-adjusted α level 0.017, pairwise comparisons between implant groups). Repeated measures ANOVA. Mixed models, repeated measures within subject. Implant type/site/configuration independent variables (length covariate). (B/SW/SC lengths compared with Kruskal-Wallis test); Test type: Equivalence — Intraclass Correlation Coefficient (ICC, two-way mixed-effect model) assessed inter- and intra-examiner reliability of bone level measurement on 20 radiographs. Dahlberg measurement error. Two-way, mixed effect model; p < 0.05, ANOVA — Bonferroni correction was applied for pairwise comparisons; Repeated measures ANOVA. Dahlberg measurement error; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.22 to -0.49], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: All Participants (Configurations 1, 2, and 3); Total 36 Swede-Vent® implants analyzed for all Configurations. Size difference expected 0.95 bone level change between B/SW/SC. Sample size 16 participants ensured 80% power to reject null hypothesis (two-sided Bonferroni-adjusted α level 0.017, pairwise comparisons between implant groups). Repeated measures ANOVA. Mixed models, repeated measures within subject. Implant type/site/configuration independent variables (length covariate). (B/SW/SC lengths compared with Kruskal-Wallis test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — Bonferroni correction was applied for pairwise comparisons; Repeated measures ANOVA. Dahlberg measurement error; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.35 to -0.64], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: All Participants (Configurations 1, 2, and 3); Total 36 Screw-Vent® implants analyzed for all Configurations. Size difference expected 0.95 bone level change between B/SW/SC. Sample size 16 participants ensured 80% power to reject null hypothesis (two-sided Bonferroni-adjusted α level 0.017, pairwise comparisons between implant groups). Repeated measures ANOVA. Mixed models, repeated measures within subject. Implant type/site/configuration independent variables (length covariate). (B/SW/SC lengths compared with Kruskal-Wallis test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — Bonferroni correction was applied for pairwise comparisons; Repeated measures ANOVA. Dahlberg measurement error; Median Difference (Final Values) = -1.77, 95% CI 2-sided [-2.13 to -1.41], Standard Error of Mean 0.18

2. Secondary Outcome: Comparison of Prosthesis, Abutment, and Implant Mobility or Looseness: Absence (0) or Presence (1) of Mobility or Looseness After 25 Years of Function
Description: Mobility was measured by applying manual pressure on the handles of two instruments, each placed on opposite sides of the prostheses and abutments, and was recorded as 0 (no mobility or looseness) or 1 (mobility or looseness). Values (Mean ± SE) were calculated, recorded and compared between B and SW, between B and SC and between SW and SC for Configuration 1 (Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1), Configuration 2 (Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2), and Configuration 3 (Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2)
Time Frame: After 25 years (24.6 ± 0.19 years, mean ± SE) of function
Population: 22 participants in all Configurations contributed 110 implants (B=36, SW=38, SC=36). One implant (B Configuration 1) had fractured; two (B and SW Configuration 2) had technical issues. 107 implants were analysed after 25 years of function. Values (Mean ± SE) were calculated, recorded and compared between all B and all SW, between all B and all SC and between all SW and all SC implant units in all three Configurations
Measure: Number; unit: Implants
Units Other Than Participants: Implants
Arm/Group | All Participants (Configurations 1, 2, and 3)
Number analyzed (Participants) | 22
Number analyzed (Implants) | 107
Implants
  Total 35 Brånemark® implants analyzed for all 3 Configurations: number analyzed (Implants) | 35
  Total 35 Brånemark® implants analyzed for all 3 Configurations | 0
  Total 36 Swede-Vent® implants analyzed for all 3 Configurations: number analyzed (Implants) | 36
  Total 36 Swede-Vent® implants analyzed for all 3 Configurations | 0
  Total 36 Screw-Vent® implants analyzed for all 3 Configurations.: number analyzed (Implants) | 36
  Total 36 Screw-Vent® implants analyzed for all 3 Configurations. | 0

3. Secondary Outcome: Comparison of Soft Tissue Healing: Height (mm) of Keratinized Tissue After 25 Years of Function
Description: Height of the keratinized tissue was measured (mm) using a ColorVue UNC12 Hu-Friedy probe on the buccal and lingual implant/abutment surfaces. Values (Mean ± SE) were calculated, recorded and compared between B and SW, between B and SC and between SW and SC for Configuration 1 (Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1), Configuration 2 (Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2), and Configuration 3 (Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2)
Time Frame: After 25 years (24.6 ± 0.19 years, mean ± SE) of function
Population: 22 participants in all Configurations contributed 110 implants (B=36, SW=38, SC=36). One implant (B Configuration 1) had fractured; two (B and SW Configuration 2) had technical issues. 107 implants were analysed after 25 years of function. Mean (Mean ± SE) values were calculated, recorded and compared between all B and all SW, between all B and all SC and between all SW and all SC implant units in all three Configurations
Measure: Mean (Standard Error); unit: mm.
Units Other Than Participants: Implants
Arm/Group | All Participants (Configurations 1, 2, and 3)
Number analyzed (Participants) | 22
Number analyzed (Implants) | 107
mm.
  Total 35 Brånemark® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 35
  Total 35 Brånemark® dental implant units analyzed for all three Configurations | 0.67 (0.08)
  Total 36 Swede-Vent® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 36
  Total 36 Swede-Vent® dental implant units analyzed for all three Configurations | 0.51 (0.08)
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 36
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations | 0.74 (0.10)

4. Secondary Outcome: Comparison of Soft Tissue Healing: Probing Depth (mm) After 25 Years of Function
Description: Using a ColorVue UNC12 Hu-Friedy probe, probing depth was measured (mm) on the buccal, lingual, mesial and distal implant/abutment surfaces. Values (Mean ± SE) were calculated, recorded and compared between B and SW, between B and SC and between SW and SC for Configuration 1(Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1), Configuration 2 (Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2), and Configuration 3 (Brånemark® 2, Swede-Vent ®1, Screw-Vent® 2)
Time Frame: After 25 years (24.6 ± 0.19 years, mean ± SE) of function
Population: 22 participants in all Configurations contributed 110 units (B=36, SW=38, SC=36). 107 were analyzed (B=35. SW=36, SC=36). fBIC-MG was measured at mesial and distal sides of each unit after 25 years of function. Mean (Mean ± SE) values were calculated, recorded and compared between all B and all SW, between all B and all SC and between all SW and all SC dental implant units in all three Configurations
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: Implants
Arm/Group | All Participants (Configurations 1, 2, and 3)
Number analyzed (Participants) | 22
Number analyzed (Implants) | 107
mm
  Total 35 Brånemark® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 35
  Total 35 Brånemark® dental implant units analyzed for all three Configurations | 2.09 (0.14)
  Total 36 Swede-Vent® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 36
  Total 36 Swede-Vent® dental implant units analyzed for all three Configurations | 2.34 (0.18)
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations: number analyzed (Implants) | 36
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations | 2.29 (0.18)

5. Secondary Outcome: Comparison of Soft Tissue Healing: Absence (0) or Presence (1) of Plaque and/or Gingival Bleeding After 25 Years of Function
Description: Absence (0) or presence (1) of plaque and/or gingival bleeding on probing was evaluated using the dichotomous/binary plaque index (dPI) (Galgut, P. A., 1999) and bleeding index (dBI), respectively (Galgut, P.A., 1999). Values (Mean ± SE) were compared between B and SW, between B and SC and between SW and SC for Configuration 1 (Brånemark® 2, Swede-Vent® 2, Screw-Vent ®1), Configuration 2 (Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2), and Configuration 3 (Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2)
Time Frame: After 25 years (24.6 ± 0.19 years, mean ± SE) of function
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | All Participants (Configurations 1, 2, and 3)
Number analyzed (Participants) | 22
Number analyzed (Implants) | 107
score on a scale
  Total 35 Brånemark® dental implant units analyzed for all three Configurations. Plaque Mean dPI: number analyzed (Implants) | 35
  Total 35 Brånemark® dental implant units analyzed for all three Configurations. Plaque Mean dPI | 0.40 (0.06)
  Total 36 Swede-Vent® dental implant units analyzed for all three Configurations. Plaque Mean dPI: number analyzed (Implants) | 36
  Total 36 Swede-Vent® dental implant units analyzed for all three Configurations. Plaque Mean dPI | 0.42 (0.06)
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations. Plaque Mean dPI: number analyzed (Implants) | 36
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations. Plaque Mean dPI | 0.43 (0.06)
  Total 35 Brånemark® dental implant units analyzed for all three Configurations. Bleeding Mean dBI: number analyzed (Implants) | 35
  Total 35 Brånemark® dental implant units analyzed for all three Configurations. Bleeding Mean dBI | 0.48 (0.06)
  Total 36 Swede-Vent dental implant units analyzed for all three Configurations. Bleeding Mean dBI: number analyzed (Implants) | 36
  Total 36 Swede-Vent dental implant units analyzed for all three Configurations. Bleeding Mean dBI | 0.47 (0.05)
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations. Bleeding Mean dBI: number analyzed (Implants) | 36
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations. Bleeding Mean dBI | 0.44 (0.06)

6. Secondary Outcome: Comparison of Soft Tissue Healing: Absence (0) or Presence (1) of Purulent Exudate After 25 Years of Function
Description: Absence (0) or presence (1) of purulent exudate on probing was evaluated. Values (Mean ± SE) were recorded, and compared between B and SW, between B and SC and between SW and SC for Configuration 1 (Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1), Configuration 2 (Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2), and Configuration 3 (Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2)
Time Frame: After 25 years (24.6 ± 0.19 years, mean ± SE) of function
Population: as for outcome 4
Measure: Number; unit: Implants.
Units Other Than Participants: Implants.
Arm/Group | All Participants (Configurations 1, 2, and 3)
Number analyzed (Participants) | 22
Number analyzed (Implants.) | 107
Implants.
  Total 35 Brånemark® dental implant units analyzed for all three Configurations. Purulent exudate: number analyzed (Implants.) | 35
  Total 35 Brånemark® dental implant units analyzed for all three Configurations. Purulent exudate | 0
  Total 36 Swede-Vent dental implant units analyzed for all three Configurations. Purulent exudate: number analyzed (Implants.) | 36
  Total 36 Swede-Vent dental implant units analyzed for all three Configurations. Purulent exudate | 1
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations. Purulent exudate: number analyzed (Implants.) | 36
  Total 36 Screw-Vent® dental implant units analyzed for all three Configurations. Purulent exudate | 0

7. Other Pre Specified Outcome: Comparison of Two Measurement Systems Used to Evaluate Peri-implant Bone Healing After 25 Years of Function
Description: Conventional peri-apical radiology and phosphor-plate digital technology (Digora System™, Digora OptimeTM, Sporedex Dental Co., Tuusula, Finland) were used with the standardized equipment to take peri-apical radiographs on 95 implant/abutment units (Camarda, et al., 2018; Bhaskaran, et al., 2005). Following calibration, the distance between the first-bone-to-implant-contact-point and the crestal-microgap (fBIC-MG) was measured (mm) at the mesial and distal aspects of each implant/abutment unit after 25 years of function. Values (Mean ± SE) fBIC-MG were recorded for each of the two measurement systems. ICC (Intraclass Correlation Coefficient, two-way, mixed effect model) and Bland-Altman Limits of agreement (Bland & Altman, 1986) were used to evaluate the level of agreement between the two systems
Time Frame: After 25 years (24.6 ± 0.19 years, mean ± SE) of function
Population: Each of the 22 participants contributed five implants for a total of 110 B=36, SW=38, SC=36) for all three configurations. However, only 95 implants (19 participants) were analyzed (B=32, SW=32, SC=31) for all three configurations in order to compare the two measurement systems. One implant (SW, Configuration 1) was fractured. Two implants (one B and one SW, both Configuration 2) had technical issues with radiographs. Twelve implants could not be measured due to participant refusal
Measure: Mean (95% Confidence Interval); unit: Implants
Units Other Than Participants: Implants
Arm/Group | All Participants (Configurations 1, 2, and 3)
Number analyzed (Participants) | 22
Number analyzed (Implants) | 95
Implants
  ICC (Intraclass Correlation Coefficient two-way, mixed effect model) | 0.93 [0.89 to 0.95]
  Bland-Altman Limits of agreement (Bland & Altman,1986) | 0.15 [-1.21 to 1.51]

ADVERSE EVENTS:
Time Frame: After 25 years (24.6 ± 0.19 years, mean ± SE) of function.
Description: All B,SW, and SC units (implants) surgically placed in participants' jaws, and restored with prostheses, at start of original project (ClinicalTrials.gov ID No. NCT01641198) 25 years previously have no possible adverse effects on the overall health of participants. B, SW, and SC implants were and remain FDA and Health and Welfare Canada approved, and have been and continue to be sold to this day internationally, with the exception of SW (Swede-Vent®) that has been discontinued.
Groups:
- Active Comparator: Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1 (Configuration 1).: Device: Brånemark® implant placed at sites 2 (left medial) and 5 (right distal), Swede-Vent® implant placed at sites 1 (left distal) and 4 (right medial), Screw-Vent® implant placed at site 3 (para symphysis).
- Experimental: Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2 (Configuration 2).: Device: Brånemark® implant placed at site 3 (para symphysis), Swede-Vent® implant placed at sites 2 (left medial) and 5 (right distal), Screw-Vent® implant placed at sites 1 O(left distal) and 4 (right medial).
- Experimental: Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3).: Device: Brånemark® implant placed at sites 1 (left distal) and 4 (right medial), Swede-Vent® implant placed at site 3 (para symphysis), Screw-Vent® implant placed at sites 2 (left medial) and 5 (right distal).
Arm/Group | Active Comparator: Brånemark® 2, Swede-Vent® 2, Screw-Vent® 1 (Configuration 1). | Experimental: Brånemark® 1, Swede-Vent® 2, Screw-Vent® 2 (Configuration 2). | Experimental: Brånemark® 2, Swede-Vent® 1, Screw-Vent® 2 (Configuration 3).
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/6

LIMITATIONS AND CAVEATS:
Study results are applicable to implants placed between mental foramena in edentulous mandibles of patients, and restored with complete prostheses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT03862482/Prot_SAP_001.pdf